CLINICAL TRIAL: NCT01765270
Title: Mechanistic Assessment of the Properties of Saxagliptin in Subjects Undergoing Coronary Artery Bypass Graft Surgery: a Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Mechanistic Assessment of the Properties of Saxagliptin in Subjects Undergoing Coronary Artery Bypass Graft Surgery
Acronym: MAPSS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to poor enrollment.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Pro00041744
Record Dates: First submitted 2013-01-04; First posted 2013-01-10 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease
Keywords: Diabetes; Diabetes Mellitus; Type 2 Diabetes; Cardiovascular Disease; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin (Active Comparator): Treatments to be administered are saxagliptin 5 mg (once daily) to begin at randomization 5 to 7 days before CABG surgery, continuing through the peri-CABG surgery period and discharge, and for a total of 30 (± 5) days post-CABG surgery.
  Interventions: Drug: Saxagliptin
- Placebo (Placebo Comparator): Treatments to be administered are placebo 5 mg (once daily) to begin at randomization 5 to 7 days before CABG surgery, continuing through the peri-CABG surgery period and discharge, and for a total of 30 (± 5) days post-CABG surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — one 5-mg saxagliptin tablet daily
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Placebo — 5mg placebo tablet daily
  Arms: Placebo

SUMMARY:
Individuals with type 2 diabetes mellitus (T2DM) are at increased risk for cardiovascular events (for example, heart attack) and the risk is related to one's overall control of blood glucose levels. In this study the investigators will measure the effects of saxagliptin, compared to placebo, before, during, and after coronary artery bypass graft (CABG) surgery. The investigators will use samples of the patients' blood and tissue to measure and evaluate indicators of the body's response to the treatment. This study is being done to evaluate the effect of saxagliptin on biomarkers of the heart to help us understand whether reducing or controlling a person's blood glucose levels during and after CABG surgery will produce better clinical outcomes (for example, better heart health).

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial to evaluate the effect of saxagliptin on cardiac biomarkers of myocardial necrosis, cardiac function, inflammation, and apoptosis in subjects with Type 2 diabetes mellitus (T2DM) undergoing CABG surgery (on pump, via a median sternotomy approach) as an integrated measure of the potential mechanistic effects of saxagliptin on prevention of cardiovascular (CV) outcomes. Approximately 74 subjects will be randomized and complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of type 2 diabetes mellitus (T2DM) with glycosylated hemoglobin (HbA1c) between 6.5% and 10%, inclusive.

  * Stable doses of oral antihyperglycemic agents for at least 2 months
  * Stable dose of chronic insulin therapy for at least 2 months
  * HbA1c documented within 3 months before study enrollment
* Planned first elective coronary artery bypass graft (CABG) surgery

Exclusion Criteria:

* Elevated Creatine Kinase-Myocardial Bands (CK-MB) or troponin level above the 99th percentile at screening
* Receiving incretin therapy or having received incretin therapy within the previous 2 months
* Type 1 DM or a history of ketoacidosis
* Women who are pregnant or breastfeeding
* Known end-stage Kidney disease
* Known sensitivity or intolerance to saxagliptin or dipeptidyl peptidase-4 (DPP-4) inhibitor
* Clinically apparent liver disease
* History of pancreatitis

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Kristin Newby, M.D., MHS, Principal Investigator — Duke University
Locations (10):
- United States (10):
  - Cardiology, PC, Birmingham, Alabama
  - Cardio-Thoracic Surgeons PC, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Stanford University Medical Center, Palo Alto, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Chippenham Medical Center, Richmond, Virginia
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin: Treatments to be administered are saxagliptin 5 mg (once daily) to begin at randomization 5 to 7 days before coronary artery bypass graft (CABG) surgery, continuing through the peri-CABG surgery period and discharge, and for a total of 30 (± 5) days post-CABG surgery.
- Placebo: Treatments to be administered are placebo 5 mg (once daily) to begin at randomization 5 to 7 days before coronary artery bypass graft (CABG) surgery, continuing through the peri-CABG surgery period and discharge, and for a total of 30 (± 5) days post-CABG surgery.
Period: Overall Study
Arm/Group | Saxagliptin | Placebo
Started | 5 | 7
Completed | 4 | 6
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population: all subjects randomized who received at least one dose of study drug (Saxagliptin or placebo) before CABG surgery and underwent a CABG, as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin | Placebo | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (5.3) | 60.2 (8.1) | 59.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Troponin I (TnI) Area Under the Curve (AUC)
Time Frame: pre-CABG surgery (after 5 to 7 days of assigned treatment, predischarge or 5 days post-CABG surgery (Approximately 12 days)
Measure: Median (Inter-Quartile Range); unit: ng*hr/mL
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
ng*hr/mL | 463.25 [228.74 to 928.29] | 235.98 [230.03 to 266.01]

2. Secondary Outcome: High Sensitive Troponin-I (hsTnT) Area Under the Curve
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng*hr/mL
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
ng*hr/mL | 213.82 [114.09 to 265.03] | 129.14 [58.25 to 181.61]

3. Secondary Outcome: Creatine Kinase-Myocardial Bands (CK-MB) Area Under the Curve
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng*hr/mL
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
ng*hr/mL | 1174.9 [1057.36 to 1301.66] | 835.76 [744.84 to 885.81]

4. Secondary Outcome: Number of Major Adverse Cardiac Events (MACE)
Description: Death, myocardial infarction (MI), or New congestive heart failure (CHF)
Time Frame: Baseline to end of study (Approximately 35-37 days)
Measure: Number; unit: Cardiac Events
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
Cardiac Events | 0 | 0

5. Secondary Outcome: Duration of Inotropic Support
Time Frame: CABG surg until hosp discharge (Approximately 5 days)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
hours | 25.67 (23.58) | 8.49 (7.60)

6. Secondary Outcome: Number of Participants Who Had an Episode of Hypoglycemia
Time Frame: baseline to end of study (Approximately 35-37 days)
Measure: Number; unit: participants
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
participants | 0 | 0

7. Secondary Outcome: Number of Participants Who Required Intraaortic Balloon Pump (IABP) Support
Time Frame: CABG to hospital discharge (Approximately 5 days)
Measure: Number; unit: participants
Groups:
- Saxagliptin: Treatments to be administered are saxagliptin 5 mg (once daily) to begin at randomization 5 to 7 days before CABG surgery, continuing through the peri-CABG surgery period and discharge, and for a total of 30 (± 5) days post-CABG surgery.daily
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
participants | 0 | 0

8. Secondary Outcome: Need for Antiarrhythmic Therapy
Time Frame: CABG surg to hospital discharge Approximately 5 days
Measure: Number; unit: participants
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 6
participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Participants were followed for aproximately 35 days (5 days before CABG and typically 30 days after CABG).
Arm/Group | Saxagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/4 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin (N=4) | Placebo (N=6)
atrial fibrillation (Cardiac disorders) | 1 | 1
Pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subject analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No